CLINICAL TRIAL: NCT03232931
Title: Randomized Controlled Trial to Improve Multisensory Neural Processing, Language & Motor Outcomes in Preterm Infants
Brief Title: Trial to Improve Multisensory Neural Processing, Language & Motor Outcomes in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Nathalie Maitre, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003034; R01HD093706 (NIH); IRB17-00025/IRB18-00579 (Other: Nationwide Children's Hospital)
Record Dates: First submitted 2017-02-03; First posted 2017-07-28 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Preterm Infant
Keywords: auditory; tactile; mother's voice; multisensory
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial design with intent-to-treat analysis in hospitalized preterm infants between 32 and 36 weeks post-menstrual age. Both the control and intervention groups will receive routine neonatal intensive care protocols (including skin-to-skin care by parent when available and daily sessions of exposure to recorded parent's voice). In addition to routine care, the parent-supported multisensory intervention consists of 10 sessions of standardized, therapist-administered, auditory-tactile stimulation that combines contingent recorded mother's voice delivered using a pacifier-activated system, during holding with supportive tactile containment against the therapist's chest, covered by cloth imprinted with mother's scent. Possible covariates, multi- and uni- sensory processing, will be measured at entry into the study and immediately after the treatment phase. Sensory reactivity will be measured at 1 year and language and motor outcomes will be assessed at 2 years.
Who Masked: Outcomes Assessor
Masking Description: Except for parent reports, all measures will be administered by masked examiners.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Multisensory Intervention (Experimental): Preterm infants in the NICU who are randomized to receive a multisensory intervention, in addition to the standard of care. The multisensory intervention uses recordings of the parents' voices and nurturing touch administered in the NICU during 12 to 23 sessions of standardized, therapist-administered, auditory-tactile stimulation, dispersed over a 2 to 3 week period. The intervention includes 2 components: (1) holding and light pressure containment of the infant against the hospital-gown covered chest of the therapist for tactile and non-specific auditory stimulation simultaneous with (2) playing of mother's voice contingent on infant pacifier sucking. Additionally, a gauze square scented with parent's skin will be used to provide olfactory stimulation.
  Interventions: Behavioral: Therapist skin-to-skin Care; Device: Contingent parent's voice exposure; Behavioral: Parental skin-to-skin care; Device: Recorded parent's voice
- Standard of Care (Other): Preterm infants in the NICU who are randomized to receive the standard of care. The standard care for preterm infants in the NICU currently follows medical protocols of skin-to-skin holding and exposure to recordings of parent's voice.
  Interventions: Behavioral: Parental skin-to-skin care; Device: Recorded parent's voice

INTERVENTIONS:
Behavioral: Therapist skin-to-skin Care — Skin-to-skin (STS) holding is part of the multisensory intervention where the therapist will wear a clean 100% cotton T-shirt with a clean hospital gown on top of the shirt and wrap the "kangaroo" positioner securely over the gown. A gauze square scented with parent's skin will be used to provide olfactory stimulation. Therapist STS sessions occur with simultaneous playing of mother's voice contingent on infant pacifier sucking.
  Arms: Multisensory Intervention
Device: Contingent parent's voice exposure — The Pacifier Activated Lullaby® (PAL®) device, is a digital music delivery system that integrates a sensor, a pacifier routinely used in the NICU, and a receiver. It delivers a predetermined 10 seconds of recorded parent's voice singing lullabies upon detection of a suck that meets a preset pressure threshold. The original systems were modified for research use by decreasing the lower limit of activation thresholds for delivering the recording. Minimal effort is required to trigger the device. However, the settings ensure that regular attempts are needed to continue to receive continual presentation of the recording of mother's voice by requiring another suck after 10 seconds. The auditory stimulation with PAL will be provided when the infants are still awake (i.e., at the beginning of the session).
  Other Names: Pacifier Activated Lullaby® (PAL®)
  Arms: Multisensory Intervention
Behavioral: Parental skin-to-skin care — The standard of care includes parental skin-to-skin care and exposure to parent's voice. During parental skin-to-skin care, infants are placed in a prone position with head positioned over the sternum, allowing transmission of breath and heart sounds to the developing ear. Deeper pressure is applied to offer support and feedback to the child's bottom. Session length is set to a minimum of 45 minutes per unit protocols.
Device: Recorded parent's voice — Per standard of care, preterm infants in the NICU currently receive noncontingent recorded parents' voice during two 20 minute sessions per day. Recordings are standardized and are played through a sterilizable device (DINO-egg).
  Other Names: DINO-egg

SUMMARY:
Every year, almost all of ½ million infants born prematurely in the US and 15 million worldwide suffer from abnormal brain maturation resulting from interactions between immaturity and atypical sensory experiences after birth. This study uses rigorous scientific methods to measure the effects and determine the mechanisms of action of a parent-supported multisensory neurorehabilitative intervention for preterm infants, adaptable to a wide variety of neonatal environments, even when parents cannot be at their child's bedside. The intervention aims to improve brain multisensory processing, reactions to sensory stimulation in the home and long term language and motor development.

DETAILED DESCRIPTION:
This study is a randomized controlled trial design with intent-to-treat analysis in hospitalized preterm infants between 32 and 36 weeks post-menstrual age. Both the control and intervention groups will receive routine neonatal intensive care unit care (i.e., skin-to-skin care by parent when available and daily sessions of exposure to recorded parent's voice). In addition to routine care, the parent-supported multisensory intervention consists of sessions of standardized, therapist-administered, auditory-tactile stimulation that combines contingent recorded mother's voice delivered using a pacifier-activated system, during holding with supportive tactile containment against the therapist's chest, covered by cloth imprinted with mother's scent. Possible covariates, multi- and uni-sensory processing, will be measured at entry into the study and immediately after the treatment phase. Event-related potential (ERP) testing will be performed prior to the prior to intervention and after intervention is complete, which occurs at 36 weeks postmenstrual age (PMA) on average. ERP testing will take approximately 30 to 40 minutes. All infants will be seen at the neonatal intensive care unit (NICU) Follow-Up Program clinics at 9-12 months PMA (Year 1) and 22-24 months PMA (Year 2), where neurodevelopmental outcomes will be assessed using standardized methods.

Parents will also have the opportunity to consent separately to a secondary part to the study in which their infant would participate in one additional ERP testing session in the NICU between 34-36 weeks PMA and one additional visit to the clinical laboratory for ERP testing between 3-4 months PMA. This optional, secondary part of the study is observational only and does not influence randomization for the main trial. For the secondary part of the study, the population will be 40 of the 230 participants. All parents who are approached for the study prospectively and are randomized to control group will be asked if they would like to participate in the secondary part. Enrollment for this secondary part of the study will stop when 40 participants are reached.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization at a study location
* Postmenstrual age of 32 weeks 0 days gestation to 36 weeks 0 days gestation

Exclusion Criteria:

* Ventilation using an endotracheal tube
* Major congenital malformations
* Family history of genetic hearing loss
* Use of sedatives or seizure medications

Secondary Study Inclusion Criteria:

* Enrolled in the control group of the main study

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2025-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie L Maitre, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richard C, Jeanvoine A, Stark AR, Hague K, Kjeldsen C, Maitre NL. Randomized Trial to Increase Speech Sound Differentiation in Infants Born Preterm. J Pediatr. 2022 Feb;241:103-108.e3. doi: 10.1016/j.jpeds.2021.10.035. Epub 2021 Oct 25. PMID 34710395
- [Derived] Neel ML, Yoder P, Matusz PJ, Murray MM, Miller A, Burkhardt S, Emery L, Hague K, Pennington C, Purnell J, Lightfoot M, Maitre NL. Randomized controlled trial protocol to improve multisensory neural processing, language and motor outcomes in preterm infants. BMC Pediatr. 2019 Mar 19;19(1):81. doi: 10.1186/s12887-019-1455-1. PMID 30890132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Nationwide Children's Hospital in Columbus, Ohio, and Grady Memorial Hospital and Emory University Hospital Midtown in Atlanta, Georgia, USA. Participant enrollment began October 29, 2018 and data collection for the assessments occurring at up to 42 weeks gestational age was completed by February 20, 2023.
Groups:
- Multisensory Intervention: Preterm infants in the neonatal intensive care unit (NICU) randomized to receive a multisensory intervention, in addition to the standard of care. The multisensory intervention uses recordings of the parents' voices and nurturing touch administered in the NICU during 12 to 23 sessions of standardized, therapist-administered, auditory-tactile stimulation, dispersed over a 2 to 3 week period. The intervention includes 2 components: (1) holding and light pressure containment of the infant against the hospital-gown covered chest of the therapist for tactile and non-specific auditory stimulation simultaneous with (2) playing of mother's voice contingent on infant pacifier sucking. Additionally, a gauze square scented with parent's skin will be used to provide olfactory stimulation.
- Standard of Care: Preterm infants in the NICU randomized to receive the standard of care. The standard care for preterm infants in the NICU currently follows medical protocols of skin-to-skin holding and exposure to recordings of parent's voice.
Period: Overall Study
Arm/Group | Multisensory Intervention | Standard of Care
Started | 126 | 122
Completed (Completed the NICU portion of the study lasting up to 42 weeks gestational age.) | 112 | 116
Not Completed | 14 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Discharged before completing study activities per protocol | 4 | 2
Not completed — Parent did not record voice | 1 | 2
Not completed — Research and staffing limitations during the Coronavirus Disease 2019 (COVID-19) pandemic | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis includes participants who completed the trial up to 42 weeks gestational age.
Groups:
- Multisensory Intervention: Preterm infants in the NICU randomized to receive a multisensory intervention, in addition to the standard of care. The multisensory intervention uses recordings of the parents' voices and nurturing touch administered in the NICU during 12 to 23 sessions of standardized, therapist-administered, auditory-tactile stimulation, dispersed over a 2 to 3 week period. The intervention includes 2 components: (1) holding and light pressure containment of the infant against the hospital-gown covered chest of the therapist for tactile and non-specific auditory stimulation simultaneous with (2) playing of mother's voice contingent on infant pacifier sucking. Additionally, a gauze square scented with parent's skin will be used to provide olfactory stimulation.
- Total: Total of all reporting groups
Arm/Group | Multisensory Intervention | Standard of Care | Total
Number analyzed (Participants) | 112 | 116 | 228
Age, Continuous [Mean (Standard Deviation); unit: Weeks postmenstrual age (PMA)] | 34.22 (1.22) | 34.14 (1.18) | 34.18 (1.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 61 | 117
  Male | 56 | 55 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 109 | 113 | 222
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 56 | 106
  White | 50 | 55 | 105
  More than one race | 9 | 1 | 10
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 116 | 228
Gestational age at birth [Mean (Standard Deviation); unit: Weeks postmenstrual age (PMA)] | 28.84 (2.79) | 28.81 (2.91) | 28.82 (2.85)

OUTCOME MEASURES:

1. Primary Outcome: Index of Multisensory Processing (IMP)
Description: Cortical processing is measured as the percentage of time spent in Event Related Potential (ERP) response patterns that have been previously characterized as typical in healthy infants born at full term. ERP is assessed through high-density functional electroencephalogram (EEG) in the NICU. The Index of Multisensory Processing (IMP) is calculated as the percentage of time that the topographical pattern of the participant's ERP to multisensory stimuli is most like template map of a full term infant. The IMP is expressed as a percentage from 100% (samples show nearly-typical activation all of the time) to 0% (samples show nearly-typical activation none of the time).
Time Frame: At enrollment up to 36 weeks gestation (prior to intervention), and at intervention completion up to 42 weeks gestation
Population: This analysis includes participants who completed the study and had analyzable event related potential (ERP) data for both study time points. ERP data were not collected for 9 participants in the Multisensory Intervention group and 10 participants in the Standard of Care group. ERP data were collected were not analyzable for 5 participants in the Multisensory Intervention group.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Multisensory Intervention | Standard of Care
Number analyzed (Participants) | 98 | 105
percentage of time
  Prior to the intervention | 31.4 (47) | 49.0 (48)
  After the intervention | 35.6 (47) | 18.8 (37)

2. Secondary Outcome: Infant/Toddler Sensory Profile (ITSP) Score
Description: The Infant/Toddler Sensory Profile (ITSP), for ages 7 to 36 months, is a 48-item questionnaire, completed by caregivers, and is used to measure sensory reactivity and adaptation to the environment. The ITSP assesses five sensory processing sections (Auditory, Visual, Tactile, Vestibular, and Oral Sensory Processing) and a General measure. Responses are given on a 5-point scale where 1 = almost always and 5 = almost never. For children 7 to 36 months there are four quadrant scores and one combined quadrant score available. For children 12 months corrected age, the four quadrant score ranges are as follows:
  Low Registration: 11-55 (typical performance is 46-54) Sensation Seeking: 14-70 (typical performance is 19-35) Sensory Sensitivity: 11-55 (typical performance is 41-52) Sensation Avoiding: 12-60 (typical performance is 45-56) Low Threshold (combined quadrant score): 23-115 (typical performance is 87-107)
Time Frame: at 12 months corrected age
Reporting Status: Not Posted

3. Secondary Outcome: Change in Bayley Scales of Infant and Toddler Development - 3rd Edition (Bayley III) Score
Description: The Bayley-III is a standardized comprehensive assessment tool for assessing child development in children one month to 42 months old. The highest possible scaled score on each subtest is 19, and the lowest possible score is 1. Scores from 8 to 12 are considered average. Composite scores for motor and language domains are derived from sums of the subtest scaled scores. Composite scores range from 40-160.
Time Frame: 12 and 24 months corrected age
Reporting Status: Not Posted

4. Secondary Outcome: Change in Preschool Language Scales - 5th Edition (PLS-5) Score
Description: The PLS-5 is a language assessment tool administered by a trained professional in which children point or verbally respond to pictures or objects. It assesses both receptive (auditory comprehension) and expressive language skills in young children, and a total language score is also calculated. Total scores for Auditory Comprehension, Expressive Communication, and Total Language are standardized with a mean of 100 and a standard deviation of 15. Scores below 100 indicate below average performance while scores above 100 indicate better than average performance.
Time Frame: 2 Years (22-26 months corrected age)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and is continuing through the final assessment at Year 2 (22-26 months corrected age).
Arm/Group | Multisensory Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/126 | 1/122
Serious Adverse Events (participants affected / at risk) | 0/126 | 1/122
Other Adverse Events (participants affected / at risk) | 6/126 | 1/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multisensory Intervention (N=126) | Standard of Care (N=122)
Hospital admission due to respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Hospitalization occurred after NICU discharge and before the 9-12 month follow-up.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multisensory Intervention (N=126) | Standard of Care (N=122)
Participant needed resuscitation measures while in NICU (Surgical and medical procedures) | 2 | 1 — Not study related
Multiple mild bradycardia/desaturation events during a session, while in NICU (Cardiac disorders) | 2 | 0 — Possibly related to the study intervention
Major event needing vigorous stimulation and free flow oxygen (blow by) to resolve, while in NICU (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Not study related
Emergency department visit for respiratory distress due to respiratory syncytial virus (RSV) (Infections and infestations) | 1 | 0 — After NICU discharge, before 9-12 month follow-up; not study related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT03232931/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03232931/ICF_000.pdf